CLINICAL TRIAL: NCT03097640
Title: Understanding Perspectives of Frequently-Admitted Hospital Patients
Acronym: CHAMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Bruce Lowell Henschen, Assistant Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: STU00203847
Record Dates: First submitted 2017-03-27; First posted 2017-03-31 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-10

CONDITIONS: Continuity of Patient Care; High Utilizers of Hospital Care; Patient-Centered Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CHAMP (Experimental): Participants enrolled in CHAMP are followed by a team of a social worker and physician across the care continuum. CHAMP team members visit patients in the ED and on inpatient floors. Along with the patient's input, the team develops an Individualized Care Plan outlining the patient's medical and social history and providing recommendations to other providers on specific aspects of their care. Care plans are reviewed with patients on an individual basis and reviewed periodically by the CHAMP providers. CHAMP-enrolled participants are scheduled for physician and social worker follow-up appointments at the CHAMP clinic; this time is used to provide intensive case management, medical care, and psychosocial support.
  Interventions: Other: CHAMP
- Standard Care (No Intervention): Individuals in the standard care arm will receive care as they do normally when hospitalized, including medical and inpatient social work services, as well as outpatient care from their providers.

INTERVENTIONS:
Other: CHAMP — CHAMP team members visit patients in the ED and on inpatient floors. Along with the patient's input, the team develops an Individualized Care Plan outlining the patient's medical and social history and providing recommendations to other providers on specific aspects of their care. Care plans are reviewed with patients on an individual basis and reviewed periodically by the CHAMP providers. CHAMP-enrolled participants are scheduled for physician and social worker follow-up appointments at the CHAMP clinic; this time is used to provide intensive case management, medical care, and psychosocial support.
  Arms: CHAMP

SUMMARY:
This study evaluates the clinical outcomes of a novel program designed to target patients who are high-utilizers of hospital services. Patients who are frequently admitted to medical services - "high-utilizers" - present a unique set of challenges to providers and the health care system that require a different way of approaching chronic illness. The Complex High Admission Management Program (CHAMP) is an innovative model of care consisting of a small team of providers who establish continuity relationships with high-utilizer patients. CHAMP strives to provide effective, high value care via a longitudinal relationship-based care model through provider continuity, intensive case management, and personalized care plans. To better understand the potential outcomes of CHAMP, this study is a longitudinal, prospective, randomized, controlled trial of medical high-utilizers enrolled in CHAMP compared to a group of high-utilizer patients receiving usual care.

DETAILED DESCRIPTION:
Frequent users of hospital services, otherwise known as hospital "high-utilizers," comprise a diverse patient population that pose unique challenges to the current US health care delivery model. The Complex High Admission Management Program (CHAMP), implemented at Northwestern Memorial Hospital in Chicago, IL, seeks to improve care for high-utilizer patients through provider continuity, intensive case management, and developing personalized care plans that span inpatient, outpatient, and emergency care environments.

Preliminary evaluation of CHAMP has shown a 38% decrease in 30-day unplanned hospital readmissions and an 18% decrease in ED encounters over a 6-month time period, when compared to an equal time period pre-CHAMP.

Patients are eligible for the program if they are readmitted to the hospital three times within a twelve-month period. Due to the time and resource limitations of the CHAMP team, not all patients meeting these criteria can be enrolled at once. Patients will thus be randomly selected to be enrolled in CHAMP or will receive usual care. This study plans to evaluate the difference in outcomes between patients enrolled in CHAMP and those receiving usual care by answering the following questions:

To what extent do high-utilizer patients enrolled in CHAMP differ in their level of trust in providers, self-assessed coping skills, daily symptom burden, perceived functionality, and attitudes about the healthcare system when compared to a control group of high utilizer patients receiving usual care? We will assess patient responses to a series of surveys assessing trust, feelings of discrimination, activation, satisfaction with care, and level of social functioning.

What are the healthcare utilization rates of high-utilizer patients enrolled in CHAMP compared to a control group of high-utilizer patients receiving usual care? We will compare rates of (a) hospital admission and (b) utilization (including length of stay) among high-utilizer patients enrolled in CHAMP as compared to high-utilizer patients not enrolled in the program.

ELIGIBILITY:
Inclusion criteria:

* Adults (18 yrs of age or older) who are admitted to Northwestern Memorial Hospital (NMH) and identified by EDW search as having two unplanned 30-day inpatient readmissions to NMH within the prior 12 months with one of two additional criteria:at least 1 readmission in the last 6 months, or a referral from one of that patient's medical providers.
* Admission to NMH during the study period (October 1, 2016 to September 30, 2018) and meeting criteria described above for CHAMP
* Ability to consent for this study (including ability to read materials printed in English, understanding and communicating in English, and able to understand the risks and benefits of participating in the study).

Exclusion Criteria:

* Patients who are admitted to the Intensive Care Unit, patients admitted to Oncology services (as we have found that this latter group has a multidisciplinary care team already in place), or patients actively followed by the Heart Failure Bridge and Transition (BAT) Team, a different quality improvement intervention designed to reduce readmissions among patients admitted for acute decompensated heart failure.
* Participants will be excluded if they are disoriented to person, place, or time, or are unable to consent for any other reason.
* Minors, pregnant women, and prisoners will also be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2020-07 (Actual); Study Completion 2021-10 (Actual)

PRIMARY OUTCOMES:
Readmission Rate | 180-days from indexed hospital discharge
  180-day Inpatient Readmission Rate (as defined by Medicare) to Northwestern Memorial Hospital

SECONDARY OUTCOMES:
Readmission Rate | 30 days from indexed hospital discharge
  Inpatient Readmission Rate
Readmission Rate | 90 days from indexed hospital discharge
  Inpatient Readmission Rate
Inpatient Admissions | 30 days from indexed hospital discharge
  Inpatient Admission Rate to Northwestern Memorial Hospital
Inpatient Admissions | 90 days from indexed hospital discharge
  Inpatient Admission Rate to Northwestern Memorial Hospital
Inpatient Admissions | 180 days from indexed hospital discharge
  Inpatient Admission Rate to Northwestern Memorial Hospital
Inpatient Admissions-total | 30 days from indexed hospital discharge
  Inpatient Admissions to all hospitals, as reported by patient
Inpatient Admissions-total | 90 days from indexed hospital discharge
  Inpatient Admissions to all hospitals, as reported by patient
Inpatient Admissions-total | 180 days from indexed hospital discharge
  Inpatient Admissions to all hospitals, as reported by patient
ER Admissions | 180 days from indexed hospital discharge
  ER Visits to Northwestern Memoria
ER Admissions | 30 days from indexed hospital discharge
  ER Visits to Northwestern Memoria
ER Admissions | 90 days from indexed hospital discharge
  ER Visits to Northwestern Memoria
ER Admissions-total | 30 days from indexed hospital discharge
  ER Visits to all hospitals, as reported by patient
ER Admissions-total | 90 days from indexed hospital discharge
  ER Visits to all hospitals, as reported by patient
ER Admissions-total | 180 days from indexed hospital discharge
  ER Visits to all hospitals, as reported by patient
Hospital Length of Stay | 180 days from indexed hospital discharge
  Average Length of Stay at NMH during time period
Hospital Length of Stay | 30 days from indexed hospital discharge
  Average Length of Stay at NMH during time period
Hospital Length of Stay | 90 days from indexed hospital discharge
  Average Length of Stay at NMH during time period
Clinic Visits | 180 days from indexed hospital discharge
  Number of total clinic visits
Patient-Centered Outcomes | 30 days from indexed hospital discharge
  Responses to PROMIS Profile Scales, Trust in Physicians, Patient Activation, and Feelings of Discrimination
Patient-Centered Outcomes | 90 days from indexed hospital discharge
  Responses to PROMIS Profile Scales, Trust in Physicians, Patient Activation, and Feelings of Discrimination
Patient-Centered Outcomes | 180 days from indexed hospital discharge
  Responses to PROMIS Profile Scales, Trust in Physicians, Patient Activation, and Feelings of Discrimination
Average costs | 180 days from indexed hospital discharge
  Estimated cost from billing code data for hospitalizations during time period

CONTACTS AND LOCATIONS:
Overall Officials: Bruce L Henschen, MD/MPH, Principal Investigator — Northwestern University Feinberg School of Medicine
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Henschen BL, Theodorou ME, Chapman M, Barra M, Toms A, Cameron KA, Zhou S, Yeh C, Lee J, O'Leary KJ. An Intensive Intervention to Reduce Readmissions for Frequently Hospitalized Patients: the CHAMP Randomized Controlled Trial. J Gen Intern Med. 2022 Jun;37(8):1877-1884. doi: 10.1007/s11606-021-07048-1. Epub 2021 Sep 1. PMID 34472021